CLINICAL TRIAL: NCT05869461
Title: Adapting an Effective Intervention for Enhancing Engagement in HIV Care to Meet the Needs of Key Populations in India
Brief Title: Improving HIV Adherence Care for Key Populations in India
Acronym: Chetana-PN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Humsafar Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01MH128162 (NIH); 1R01MH128162-01A1 (NIH)
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Treatment Adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention and assessment study staff do not overlap and all reasonable care is taken to keep assessment staff blinded to intervention allocation for the whole duration of the study. Investigators know intervention arm on a need to know basis but do not have contact with participants directly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive access to the wellness sessions that have specific content geared towards our key populations and they will also receive peer navigation for 6 months.
  Interventions: Behavioral: KP Specific Wellness Sessions; Behavioral: Peer Navigation
- Control (No Intervention): Control arm participants will receive standard HIV care through the Mumbai Districts AIDS Control Society (MDACS)-run ART clinics. In addition, participants will have access to an abbreviated version of the wellness groups to help them remain engaged with the study team and to control for attention.

INTERVENTIONS:
Behavioral: KP Specific Wellness Sessions — The sessions will include content on yoga, nutrition, legal issues, medical information, and community resources from the original Chetana intervention (further described below). They will also include expanded content informed by our previous studies and focus group discussions with MSM and TGW that addresses the needs for sessions on mental health, financial literacy, substance use, legal rights for key populations and coping skills for interacting with the legal system, and community resources for MSM and TGW. Sessions will include specifically tailored content related to the needs of MSM or TGW.
  Arms: Intervention
Behavioral: Peer Navigation — Participants will be assigned to a peer navigator (PN) who will be their principal point of contact for the intervention. Within a week, the navigator will set up an initial introductory meeting, either in person or via video chat. This will serve as the first monthly check-in to monitor a participant's progress. During these in-person digital meetings, the navigator will work with a participant to identify their unique barriers that currently affect engagement in care and train participants to identify and break down solutions into manageable steps. Special attention will be paid to barriers associated with intersectional stigma and PNs will draw on their own experiences as members of stigmatized groups in identifying and brainstorming successful coping strategies. While this is not a structural intervention, PNs will work with their clients to develop ways of coping with structural barriers, including transportation and referrals to social services.
  Arms: Intervention

SUMMARY:
This study seeks to adapt and pilot test a comprehensive wellness program to address the barriers to engagement in the HIV care continuum among men who have sex with men (MSM) and transgender women (TGW) in India. The content involves an adaptation of the earlier Chetana wellness adherence intervention which was found to successfully improve adherence and viral suppression among mainstream Indian persons living with HIV (PLWH). Based on the initial formative work, the adaptation includes added wellness group content and will be offered in a flexible format. It also uses peer navigators (PN), rather than Master-level counselors, to deliver tailored support at mutually convenient times and places. This PN model has been used successfully by Indian collaborators and in previous research in South Africa to link and retain PLWH in care. The intervention is intended to break the link between stigma and care seeking, which is especially important for key populations (KPs), who must deal with historically hostile legal environments and substantial isolation that further reduces engagement in HIV preventive practices and services .

Investigators are conducting this research to address the following aims:

1) To engage community stakeholders in the adaptation and pilot testing of the Chetana-PN wellness adherence intervention for use with Indian MSM and TGW who are living with HIV and who are newly or insufficiently engaged in care.

2a) To assess in a small randomized control trial (RCT) the acceptability and feasibility of the theoretically-guided, adapted intervention and to obtain preliminary effect size estimations for the impact of the intervention on engagement in care, among MSM and TGW.

2b) To characterize participant and navigator experiences in the Chetana-PN intervention and describe the practices that were most successful at overcoming barriers to care with 25 participants who received the Chetana-PN intervention and the peer navigators. These findings will subsequently be used to inform a future RCT designed to establish the efficacy of this adapted Chetana-PN intervention for sexual minorities in India.

DETAILED DESCRIPTION:
The "Chetana-PN" study aims to improve engagement in care among two key populations living with HIV -MSM and TGW in the Indian state of Maharashtra, which has both India's highest HIV prevalence and LGBT population.

Aim 1: To engage community stakeholders in the adaptation of the Chetana-PN wellness adherence intervention for use with Indian MSM and TGW who are living with HIV. Building on the original Chetana intervention and using the steps described in the adaptation framework12, investigators will add population-specific content and a peer navigator component to provide tailored support. To ensure the content fully meets MSM and TGW needs, investigators will then conduct a stakeholder workshop and incorporate their recommendations. Workshop input will be used to finalize a project manual of operations, which will be presented to stakeholders for review. Subsequently, study procedures and adapted content will be piloted with 10 participants and gather feedback to determine if additional modifications are needed to finalize.

Aim 2A: To assess in a RCT the acceptability and feasibility of the theoretically-guided, adapted intervention and obtain preliminary effect size estimations for the impact of the intervention on (1) appointment keeping, (2) ART adherence, and (3) viral suppression among MSM and TGW who are newly or insufficiently engaged in HIV care. 110 MSM and TGW living with HIV and sub-optimally engaged in care will be randomized to an acceptability and feasibility trial of the adapted Chetana-PN intervention versus a wellness attention control arm. Both groups will receive standard ART center medical treatment and counseling. Data will be collected over 12 months using interviewer-administered questionnaires, ART center booklets and viral load. Data will be analyzed to preliminarily examine whether the intervention impacts model drivers of care-seeking behaviors. These include depression, stigma, disclosure, and barriers to care.

Aim 2B: To characterize participant and navigator experiences in the Chetana-PN intervention and describe the practices that were most successful at overcoming barriers to care. 25 intervention participants and three navigators will be interviewed at the end of their involvement in the intervention to identify practices and other intervention components that were more and less successful at keeping the participants engaged in care and adherent to their ART regimens. The data will also shed additional light on the acceptability and feasibility of the intervention. Data will contextualize the findings from the pilot trial and inform a future RCT designed to establish the efficacy of Chetana-PN intervention for sexual minorities in India.

The proposed intervention adaptation builds upon the original Chetana intervention, tailoring content, enhancing flexibility, and adding a peer navigation component based on work conducted by the study team in India and other settings. The intervention involves wellness sessions with KP specific content and flexibility and peer navigation. The Control arm will receive general wellness sessions without any content focusing on engagement in care. Given the challenges of MSM and TGW to attend groups with fixed schedules, the Chetana-PN groups will be offered on a drop-in basis and scheduled at multiple times.

Participants assigned to the intervention arm will be assigned to a peer navigator who will be their principal point of contact for the intervention. The navigator will work with a participant to identify their unique barriers that currently affect engagement in care and train participants to identify and break down solutions into manageable steps. Special attention will be paid to barriers associated with intersectional stigma and PNs will draw on their own experiences as members of stigmatized groups in identifying and brainstorming successful coping strategies. While this is not a structural intervention, PNs will work with their clients to develop ways of coping with structural barriers, including transportation and referrals to social services.

Participants will be interviewed by trained study staff in a private space. Questionnaires and reviews of ART clinic booklets assessing outcome and model variables measured by our group in prior studies will be performed at BL, 6, 9 and 12 months. Responses will be entered into a tablet-based version of REDCap mobile app. REDCap is a tool used to capture and store data in a secure way. The interviews will be conducted by experienced staff members who are fluent in Hindi, Marathi and English and who will undergo training that includes interviewing techniques, standard operating procedures, human subjects protections and the study protocol.

Viral load testing will be conducted by the study at baseline and by the ART center at follow-up visits, using the same lab.

25 intervention participants (15 MSM and 10 TGW) and the navigators will be enrolled into qualitative interviews to discuss their experiences with the intervention. To ensure intervention experiences can be recalled accurately, enrollment of intervention participants for interviews will be on a rolling basis, with each selected participant being interviewed within one month of intervention completion. Navigators will be eligible for interviews after completing delivery of services to all assigned participants.

The following criteria will be used to determine if the intervention is sufficiently acceptable and feasible for an RCT: 1) Ability to recruit an average of 7 participants/week (in order to ensure enrollment of n=500 over 18 months in a future RCT); 2) Retention of at least 80% of participants with complete data; 3) All intervention participants will attend at least one monthly PN meeting or video chat and one drop-in group per month.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Speak Hindi, Marathi, or English
* Self-identify as MSM or TGW
* Be HIV-positive
* Be either newly linked to ART clinic or be insufficiently engaged in care (defined as having missed or been more than 10 days late for one clinic appointment in the past year, missed more than 10% of their pills in the past month, or have detectable viral loads after more than 6 months on ART)- Be willing and able to give informed consent.

Exclusion Criteria:

* Impaired cognitive functioning indicating potentially diminished capacity to participate in the study
* Participation in the pilot (AIM 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — MSM or TGW
Enrollment: 110 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Appointment Keeping Frequency | Baseline to 12 months
  Data on kept ART clinic appointments will be obtained from the ART clinic booklet (aka "the green book") carried by participants. This procedure has been used successfully in our previous studies with similar populations.
Change in Medication Adherence | Baseline to 12 months
  Self-report using validated self-reported measures used previously by our team with similar populations in India to assess percent of pills taken in past month and number/ days of treatment interruptions
Change in Viral Load | Baseline to 12 months
  Viral load will be tested using a validated real-time PCR assay by Metropolis laboratories, authorized and used by MDACS. The study will arrange and pay for baseline VL tests. Subsequent tests, conducted at each 6-month visit will be conducted by the ART center as part of their "Fast Track City" protocol. All analyses will be conducted by the same laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ekstrand, Ph.D, Principal Investigator — University of California; Wayne Steward, Ph.D, Principal Investigator — University of California
Locations (1):
- The Humsafar Trust, Mumbai, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data